CLINICAL TRIAL: NCT06218173
Title: Clinical Impact of Local Anaesthetic Timing on Sedation Stability and Propofol Dosage in Paediatric Dental Sedation
Brief Title: Local Anesthesia Impact on Dental Sedation
Status: Completed | Type: Observational
Sponsor: Ankara University (Other)
Responsible Party: Principal Investigator, Cagil Vural, Assoc. Prof., Ankara University
Other Study IDs: 36290600/55
Record Dates: First submitted 2024-01-12; First posted 2024-01-23 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2024-01

CONDITIONS: Sedative Overdose

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (2):
- Early LA group: The group that received LA at the induction of the sedation
- Late LA group: The group that received LA at the end of the sedation

SUMMARY:
The goal of this observational study is to investigate the impact of local anesthesia in health children who were sedated for dental procedures.

The main questions it aims to answer are:

* Impact of local anesthesia on sedation depth and hemodynamic parameters
* Impact of presence of local anesthesia on the requirement of propofol to maintain deep sedation.

Participants were deeply sedated and one group received local anesthesia at the anesthesia induction, while other group of patients received local anesthesia after the maintenance anesthesia was discontinued.

If there is a comparison group:

DETAILED DESCRIPTION:
Local anaesthesia (LA) is often preferred for stabilization of vital signs, depth of anaesthesia in dental restorations but the optimal timing of LA administration during sedation is varies according to personal preferences of dentists. Aim of this retrospective study is to investigate the effects of the timing of LA on hemodynamic parameters, depth of anaesthesia and total dose of anaesthetic drugs given in paediatric patients sedated for dental procedures.

Records of healthy children who were sedated for dental restorations will be divided into two groups. Patients who received LA at the beginning of sedation or who received LA at the end of sedation after completion of restorations. It is planned to compare the patient groups in terms of demographic data, hemodynamic data, BIS scores, Ramsey Sedation Scale scores, total propofol dose administered.

ELIGIBILITY:
Inclusion Criteria:

Paediatric dental patients who were previously sedated and fulfilled the following inclusion criteria were included in this investigation. Patients with an American Society of Anesthesiologist (ASA) physical status classification of I-II and aged between 2 and 8 years were included in the study.

Exclusion Criteria:

Exclusion criteria were ASA status III-V, age older than 8 years, having any history of allergy to anaesthetic drugs and renal disease interfering with drug metabolism.

Ages: 2 Years to 8 Years | Sex: All
Age Groups: Child
Study Population: ASA I-II pediatric patients who were deeply sedated for dental restorations in a tertiary university hospital.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
Estimate the effect of local anesthesia on sedation depth | 1 year
Estimate the effect of local anesthesia on hemodynamic parameters | 1 year
Estimate the effect of local anesthesia on total propofol requirement | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara University Faculty of Dentistry, Ankara, Turkey (Türkiye)